CLINICAL TRIAL: NCT01095887
Title: A Single Center, Open-label Study to Determine the Safety and Efficacy of a Dosing Regimen of Eculizumab Added to Conventional Treatment in the Prevention of Antibody-mediated Rejection (AMR) in ABO Blood Group Incompatible Living Donor Kidney Transplantation (ABOi LDKTx)
Brief Title: Eculizumab to Prevent Antibody-mediated Rejection in ABO Blood Group Incompatible Living Donor Kidney Transplantation
Acronym: ABOi
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Mayo Clinic (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Mark Stegall, MD, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-003392; UL1TR000135 (NIH)
Record Dates: First submitted 2010-03-26; First posted 2010-03-30 (Estimated); Results first posted 2015-06-19 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-06

CONDITIONS: Kidney Transplant
Keywords: ABO incompatibility; living donor kidney transplant; kidney transplant; ABO blood type incompatible
MeSH Terms: interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- eculizumab (Experimental): Eculizumab was given on Day 0, day 1, and weekly for the first four weeks after transplant.
  Interventions: Drug: Eculizumab

INTERVENTIONS:
Drug: Eculizumab — Subjects received eculizumab intravenously at the time of transplant, on the day after transplant, then weekly for four weeks. At four weeks post transplant, anti-blood group antibody levels were determined. Subjects may have potentially received eculizumab every two weeks for one year depending on antibody levels.
  Other Names: Soliris

SUMMARY:
The purpose of this study is to try to determine if the drug eculizumab can help prevent antibody-mediated rejection in patients undergoing a kidney transplant from a living donor with a different blood type than their own.

DETAILED DESCRIPTION:
Kidney transplantation is considered the best therapy for patients with end-stage renal disease. In some instances, the only suitable living kidney donor is ABO blood group incompatible. This usually presents a barrier to successful transplantation because most recipients have circulating serum antibodies that bind to incompatible blood groups that will bind and damage the kidney allograft early after transplantation. Fortunately, over the past decade, we and others have developed protocols involving the pretransplant removal of anti-blood group antibodies using multiple plasmapheresis treatments that allow for the successful transplantation of ABOi LDKTx. Thus, this therapy enables patients to receive a living donor with its advantages rather than having to wait >5 years for a deceased donor kidney.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Have end stage renal disease (ESRD) and is receiving a kidney transplant from a living donor to whom he/she has a baseline anti-blood group titer >1:32
* Be vaccinated against N. meningitides (quadrivalent vaccine), H. Flu, and pneumococcal disease at least two weeks prior to beginning desensitization.

Exclusion Criteria:

* Has an unstable cardiovascular condition
* Has had a previous splenectomy
* Has any active bacterial or other infection
* Has a known or suspected hereditary complement deficiency
* Has known hypersensitivity to the treatment drug or any of its excipients
* Has history of illicit drug use or alcohol abuse within the previous year
* Has history of meningococcal disease
* Has any medical condition that, in the opinion of the investigator, might interfere with the patient's participation in the study, pose an added risk for the patient, or confound the assessment of the patient (e.g. severe cardiovascular or pulmonary disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Stegall, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from May 2010 to September 2012 at the Mayo Clinic in Rochester, Minnesota.
Period: Overall Study
Arm/Group | Eculizumab
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Eculizumab
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Antibody-Mediated Rejection (AMR) Within 3 Months of Kidney Transplant
Time Frame: 3 months after kidney transplant surgery
Measure: Number; unit: participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 6
participants
  Yes | 2
  No | 4

ADVERSE EVENTS:
Time Frame: Adverse events were collected and recorded at each subject interface, up to one year after transplant.
Arm/Group | Eculizumab
Serious Adverse Events (participants affected / at risk) | 5/6
Other Adverse Events (participants affected / at risk) | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eculizumab (N=6)
Prolonged hospitalization (Cardiac disorders) | 1 (1)
Native kidney mass (Renal and urinary disorders) | 1 (1)
Native Nephrectomy (Renal and urinary disorders) | 1 (1) — Native nephrectomy due to renal mass
Partial small bowel obstruction (Gastrointestinal disorders) | 2 (2)
Elevated creatinine (Renal and urinary disorders) | 2 (2)
Splenectomy (Surgical and medical procedures) | 1 (1)
Hyperkalemia (Cardiac disorders) | 1 (1)
Elevated T- Waves (Cardiac disorders) | 1 (1)
Ogilvie's syndrome (Gastrointestinal disorders) | 1 (1)
Allograft Nephrectomy (Renal and urinary disorders) | 2 (2)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Moved to intensive care unit for 24 hours for monitoring
Antibody-mediated rejection of transplant (Renal and urinary disorders) | 2 (2)
Wound dehiscence with cecal rupture (Skin and subcutaneous tissue disorders) | 1 (1)
Right hemicolectomy (Surgical and medical procedures) | 2 (2)
Wound debridement (Surgical and medical procedures) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Platelet dysfunction (Blood and lymphatic system disorders) | 1 (1)
Thrombotic microangiopathy (Renal and urinary disorders) | 1 (1)
Pulmonary Blastomycosis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eculizumab (N=6)
Atrial Fibrillation (Cardiac disorders) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
High-volume serous drainage from surgery incision site (Surgical and medical procedures) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Lymphocele (Surgical and medical procedures) | 1 (1)
Debilitation (General disorders) | 1 (1) — Due to prolonged hospitalization

LIMITATIONS AND CAVEATS:
The study was terminated early due to poor enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes